CLINICAL TRIAL: NCT04745936
Title: Comparison of Different Stylet Angles for Orotracheal Intubation Using C-MAC® Video Laryngoscopes in Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Ji-Hyun Lee, Associate professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: H2011-196-1178
Record Dates: First submitted 2021-02-04; First posted 2021-02-09 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Intubation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- C-curve group (group C) (Experimental): In group C, stylet curvature is made similar to the natural curvature of endotracheal tube.
  Interventions: Other: Style curve similar to natural curvature of endotracheal tube
- Hockey stick curve group (group H) (Active Comparator): In group H, stylet curvature is made similar to hockey stick shape.
  Interventions: Other: Style curve similar to hockey stick shape

INTERVENTIONS:
Other: Style curve similar to natural curvature of endotracheal tube — Stylet curvature is made similar to the natural curvature of endotracheal tube for intubation using C-MAC videolaryngoscope.
  Arms: C-curve group (group C)
Other: Style curve similar to hockey stick shape — Stylet curvature is made similar to hockey stick shape for intubation using C-MAC videolaryngoscope.
  Arms: Hockey stick curve group (group H)

SUMMARY:
The purpose of this study is to investigate whether the difference in stylet curvature affects the ease of tracheal intubation using C-MAC videolaryngoscope in infants under 1 year of age.

ELIGIBILITY:
Inclusion Criteria:

① Infants under 1 year old scheduled for elective surgery under general anesthesia

② American Society of Anesthesiology physical status I, II

Exclusion Criteria:

* Any pulmonary disease

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 114 (Actual)
Dates: Start 2021-03-03 (Actual); Primary Completion 2022-05-20 (Actual); Study Completion 2022-05-20 (Actual)

PRIMARY OUTCOMES:
Tube handling time | during procedure
  From glottis visualization to completion of tracheal intubation

SECONDARY OUTCOMES:
Total intubation time | during procedure
  From insertion of C-MAC blade to completion of tracheal intubation
Time to reaching glottis | during procedure
  From visualization of glottis to reaching the glottis of tube tip
The location of the initial tube tip | during procedure
  The location of the initial tube tip on the screen of C-MAC
Successful tracheal intubation | during procedure, within 30 sec
  Incidence of successful intubation within 30 sec
Additional manipulation of stylet angle | during procedure
Number of external laryngeal manipulation | during procedure
Easiness of tracheal intubation | during procedure
  Visual analogue scale (0-10, 0: extremely easy, 10: extremely difficult)

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea